CLINICAL TRIAL: NCT01769885
Title: A Pilot Clinical Trial of Neoadjuvant Tivozanib in Localized Renal Cell Carcinoma
Brief Title: Tivozanib Before Surgery in Treating Patients With Localized Kidney Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 220412; NCI-2012-03185 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Stage II Renal Cell Cancer; Stage III Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (tivozanib and surgery) (Experimental): Patients receive tivozanib PO QD on days 1-21. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. 25 days after completion of tivozanib, patients undergo curative nephrectomy.
  Interventions: Drug: tivozanib; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: tivozanib — Given PO
  Other Names: AV-951; oral VEGF receptor tyrosine kinase inhibitor AV-951
Procedure: therapeutic conventional surgery — Undergo nephrectomy

SUMMARY:
This clinical trial studies tivozanib before surgery in treating patients with localized kidney cancer. Tivozanib may stop the growth of tumor cells by blocking some of the growth factors needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of conducting a trial of tivozanib in the neoadjuvant setting of localized (completely resectable) renal cell cancer (RCC).

SECONDARY OBJECTIVES:

I. To evaluate the safety of tivozanib in the neoadjuvant setting. II. To compare the tissue before and after tivozanib for pharmacodynamic purposes (tumor infiltrating lymphocytes, myeloid derived suppressor cells, necrosis in the primary tumor after exposure to tivozanib).

III. To assess the overall response rate of tivozanib in primary tumors and correlate the radiographic changes, if any, to histo-pathological changes in the pathology specimen post-nephrectomy.

IV. To compare the various growth factors (vascular endothelial growth factor [VEGF], interleukin-8 [IL-8], placenta growth factor [P1GF]) at baseline and post treatment.

V. To assess the nephrectomy rate after applying neoadjuvant tivozanib in this primarily resectable RCC population.

OUTLINE:

Patients receive tivozanib orally (PO) once daily (QD) on days 1-21. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. 25 days after completion of tivozanib, patients undergo curative nephrectomy.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven non-metastatic clear cell RCC, as per radiographic studies is T2 - T3a based on the American Joint Committee on Cancer (AJCC) 6th edition criteria
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Hemoglobin >= 10 gm/dL
* Absolute neutrophil count (ANC) >= 1.5 X 10^9/L
* Platelets >= 100 X 10^9/L
* Total bilirubin < 1.5 X upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 X ULN
* International normalization ratio (INR) < 1.5
* Activated partial thromboplastin time (aPTT) < 1.2 X ULN
* Serum creatinine < 1.5 mg/dL or if >= 1.5 mg/dL: calculated creatinine clearance (CrCL) > 30 mL/min based on Cockroft-Gault formula
* Must have the ability to swallow and retain oral medication
* Patients of childbearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive tivozanib (solitary kidney, multiple tumors in the same or contralateral kidney)
* Not a candidate for surgery
* Received an investigational agent within 30 days prior to enrollment
* Non-clear cell or sarcomatoid histology
* Patients with metastatic disease at presentation
* Prior therapy with tyrosine kinase inhibitor for RCC
* A second primary malignancy (except squamous and basal cell carcinoma of skin) in the past 3 years
* Active or chronic infections
* Significant cardiovascular disease, including:

  * Clinically symptomatic left ventricular failure
  * Uncontrolled hypertension: systolic blood pressure of > 150 mmHg or diastolic blood pressure of > 100 mmHg documented on 2 consecutive measurements taken at least 24 hours apart
  * Myocardial infarction, severe angina, or unstable angina within 6 months prior to administration of first dose of tivozanib
  * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation)
  * Cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication)
  * Coronary or peripheral artery bypass graft within 6 months of screening
* History of coronary artery disease or peripheral arterial disease
* History of stroke or carotid endarterectomy
* Patients who are taking cytochrome P450 system (CYP)3A4 inducers are excluded; patients taking CYP3A4 inducers that can be safely replaced with another agent may be enrolled after a 5 day washout period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03-14 (Actual); Primary Completion 2013-06-14 (Actual); Study Completion 2013-12-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting a trial of tivozanib in terms of patients completing 2 courses of tivozanib | Up to 30 days after surgery

SECONDARY OUTCOMES:
Short-term efficacy defined as a composite of presence of partial response/stable disease/complete response assessed radiographically and correlated with the nephrectomy specimen per the Response Evaluation Criteria in Solid Tumors (RECIST) criteria | Up to 30 days after surgery
  Response rate will be examined using the sample proportion and corresponding 95% confidence interval.
Incidence of adverse events evaluated using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Saby George, Principal Investigator — Roswell Park Cancer Institute